CLINICAL TRIAL: NCT05908929
Title: Comparative Evaluation of Clinical Parameters in Early-Stage III Grade A Periodontitis Patients After Insertion of Platelet Rich Fibrin as Step 2 Phase I Therapy in Periodontal Pockets: A Randomized Clinical Trial
Brief Title: PRF Therapy for Pocket Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Niccoló Giuseppe Armogida, Doctor in Dental Sciences, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/2023
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Periodontal Pocket; Periodontitis
MeSH Terms: conditions — Periodontal Pocket; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients treated with SRP and insertion of PRF (Experimental)
  Interventions: Procedure: SRP and concomitant insertion of PRF membrane
- patients treated with SRP (Active Comparator)
  Interventions: Procedure: SRP

INTERVENTIONS:
Procedure: SRP and concomitant insertion of PRF membrane — The pockets were treated with scaling and root planing (SRP) along with the simultaneous insertion of a Platelet Rich Fibrin (PRF) membrane. Blood samples were drawn without anticoagulants in 10 mL tubes, which were immediately centrifuged at 4000 rpm for 8 minutes. Upon centrifugation, the blood showed three distinct layers: the uppermost layer contained platelet poor plasma, the middle layer consisted of a fibrin clot, and the lowermost band appeared bright red due to the presence of red blood cells. The fibrin clot polymerized in a diffuse manner within the tube, which was then cut with sharp scissors and squeezed between two glass slides to obtain a thick membrane. The PRF membrane was carefully handled using a carrier and isolated with a periodontal pack dressing (Coe-Pak). All patients were followed up at one week and six weeks after the treatment.
  Arms: patients treated with SRP and insertion of PRF
Procedure: SRP — The pockets were treated using the conventional procedure of scaling and root planing (SRP) utilizing curettes and an ultrasonic device. All patients were followed up at one week and six weeks after the treatment.
  Arms: patients treated with SRP

SUMMARY:
Periodontal regenerative therapy has focused on various non-surgical and surgical treatment methods. Platelet-rich fibrin (PRF) has shown to possess multiple uses, including properties that promote healing of both soft and hard tissues. In the present study, we hypothesized that the addition of PRF into periodontal pockets, as an adjunct to conventional scaling and root planing (SRP), would enhance the outcomes of non-surgical periodontal therapy. This split-mouth randomized controlled clinical trial included 26 periodontal pocket sites in 13 patients with periodontitis. The pockets were randomly assigned as either test or control sites. In the test group, PRF was placed as an adjunct to SRP, while the control group received SRP alone. Probing pocket depths (PPD), clinical attachment levels (CAL), gingival recession (GR), plaque index (PI), and gingivitis index (GI) were measured at baseline and at six weeks. The wound healing index was measured during the six-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* either gender,
* aged 18 years or older,
* patients without a medical history of systemic diseases,
* patient with chronic periodontitis
* patient with 5 or 6 mm of probing depth

Exclusion Criteria:

* patients with medical history of systemic disease or bleeding disorders
* presence of other gingival diseases (such as leukoplakia, lichen planus, pemphigoid disorders, pemphigus vulgaris, herpetic lesions, Necrotizing Ulcerative Periodontitis (NUP)
* pregnancy
* history of any drug usage affecting the periodontium for the past six months (such as systemic antibiotic therapy)
* previous periodontal treatment in the last six months
* smoking
* teeth with untreated caries
* endodontic lesions and grade II or more mobility
* subjects with acute exacerbation of periodontitis
* patients with systemic
* disease or condition that could affect tissue healing (e.g., autoimmune disease)
* severe furcation involvement (grade II and III)
* abutment for prosthetic rehabilitation
* active orthodontic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
pocket depth | 6 weeks
  Probing pocket depths (PPD), clinical attachment levels (CAL), gingival recession (GR), plaque index (PI), and gingivitis index (GI) were measured

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Naples Federico II, Naples
  - Università degli Studi di Napoli Federico II, Napoli

IPD SHARING:
Plan to Share IPD: Undecided
There will be not necessary